CLINICAL TRIAL: NCT05590754
Title: Acute 50% Body Weight Static Axial Loading Reverses Stature Increases, Lumbar Disc Expansion and Vertebral Compliance Modulation Induced by 4 Hours of Hyper-buoyancy Floatation
Brief Title: 50% Body Weight Reverses Stature, Lumbar Disc Expansion and Vertebral Compliance by Hyper-Buoyancy Floatation.
Status: Completed | Type: Observational
Sponsor: Universidad Autonoma de Madrid (Other)
Collaborators: Centro Superior de Estudios Universitarios Lasalle (Unknown); King's College London (Other)
Responsible Party: Principal Investigator, David Marcos, Principal Investigador, Universidad Autonoma de Madrid
Other Study IDs: HR-18/19-11548
Record Dates: First submitted 2022-10-18; First posted 2022-10-21 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Intervertebral Disc Compression; Muscle Atrophy; Spine Injury
MeSH Terms: conditions — Muscular Atrophy; Spinal Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: 8 participants (4 males, 25.5±4.4 years, 63.5±10.6 kg, 163.2±5.6 cm)
  Interventions: Device: Hyper-buoyancy Floatation (HBF); Device: Axial Load after 4h of HBF
- Observational Group: 8 participants (3 males, 27.0±2.0 years, 68.4±11.8 kg, 176.5±10.9 cm
  Interventions: Device: Hyper-buoyancy Floatation (HBF); Device: Axial Load after 4h of HBF

INTERVENTIONS:
Device: Hyper-buoyancy Floatation (HBF) — Participants remained on a waterbed encased within a wooden frame partially (≈50%) filled with water super-saturated with magnesium sulphate at a temperature between 34-36°C regulated by an ultra-thin underbed heater. Participants remained supine and motionless when lay on the HBF except for temporary passive re-orientation to/and back from the prone position for vertebral compliance assessment
Device: Axial Load after 4h of HBF — Participants from observational sat upright in a chair without back support for 15 min before post testing (1G), whilst experimental group participants performed a 30s seated squat with 50% of their body weight (BW) before returning to the upright seated position.

SUMMARY:
Study with the aim to see the effect on a space ground analogue , Hyper-Buoyancy Floatation (HBF) on lumbar column and the effect of a supplementary 50% of an axial load.

DETAILED DESCRIPTION:
the aim of this study was to determine the effect of 15min of 1g reloading following 4h HBF unloading with, and without 30s of seated static 50% BW axial loading upon stature, lumbar Intervertebral Disc height (via ultrasound), vertebral compliance changes, and back pain.

ELIGIBILITY:
Inclusion Criteria:

* physical requirements (1.57-1.90m, 50-95kg)

Exclusion Criteria:

* current back/neck pain, musculoskeletal disorder, cardiovascular disease, spine surgery and being, or suspected to be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: NASA astronaut criteria (1.57-1.90m, 50-95kg)
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Height | 2 years
  Standing stature measured by a commercial stadiometer (Seca 217, Germany)

SECONDARY OUTCOMES:
Intervertebral Disc Height | 2 years
  Disc height (L2-S1) measured by ultrasound
Vertebral Stiffness | 2 years
  Vertebral stiffness from L1 to L5 was assessed passively (in the prone position) with a handheld differential vertebral compliance transducer (PulStar, Sense Technology Inc., USA) in Newtons.
Self-reported back pain | 2 years
  Pain rating scale (CHAPS) from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: David Green, PhD, Study Director — King's College London
Locations (2):
- Universidad Autónoma de Madrid, Madrid, Spain
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data is going to be shared between the investigators authors

REFERENCES:
- [Background] Swanenburg J, Langenfeld A, Easthope CA, Meier ML, Ullrich O, Schweinhardt P. Microgravity and Hypergravity Induced by Parabolic Flight Differently Affect Lumbar Spinal Stiffness. Front Physiol. 2020 Sep 2;11:562557. doi: 10.3389/fphys.2020.562557. eCollection 2020. PMID 32982803
- [Result] Green DA, Scott JPR. Spinal Health during Unloading and Reloading Associated with Spaceflight. Front Physiol. 2018 Jan 18;8:1126. doi: 10.3389/fphys.2017.01126. eCollection 2017. PMID 29403389
- [Result] Marshburn TH, Hadfield CA, Sargsyan AE, Garcia K, Ebert D, Dulchavsky SA. New heights in ultrasound: first report of spinal ultrasound from the international space station. J Emerg Med. 2014 Jan;46(1):61-70. doi: 10.1016/j.jemermed.2013.08.001. Epub 2013 Oct 15. PMID 24135505
- [Result] Chang DG, Healey RM, Snyder AJ, Sayson JV, Macias BR, Coughlin DG, Bailey JF, Parazynski SE, Lotz JC, Hargens AR. Lumbar Spine Paraspinal Muscle and Intervertebral Disc Height Changes in Astronauts After Long-Duration Spaceflight on the International Space Station. Spine (Phila Pa 1976). 2016 Dec 15;41(24):1917-1924. doi: 10.1097/BRS.0000000000001873. PMID 27779600